CLINICAL TRIAL: NCT01861015
Title: Use of Vasopressin Versus Epinephrine to Reduce Hemorrhage During Myomectomy: a Randomized Controlled Trial
Brief Title: Vasopressin Versus Epinephrine in Myomectomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CHA University (Other)
Responsible Party: Principal Investigator, Taejong Song, Professor, CHA University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KNC13-013
Record Dates: First submitted 2013-05-21; First posted 2013-05-23 (Estimated); Last update posted 2016-01-22 (Estimated); Status verified 2016-01

CONDITIONS: Uterine Myomas
MeSH Terms: interventions — Epinephrine; Vasopressins

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Epinephrine (Experimental): In the epinephrine group, we used a dilute epinephrine, 0.5 mg of epinephrine ([1/2] vial of 1mg/mL) in 50 mL of saline solution, taking care to use no more than 20 mL of solution per a subject.
  Interventions: Drug: Epinephrine
- Vasopressin (Active Comparator): In the vasopressin group, a dilute vasopressin, 5 units in 50 mL of saline solution, taking care to use no more than 20 mL of solution per a subject was injected.
  Interventions: Drug: Vasopressin

INTERVENTIONS:
Drug: Epinephrine
  Arms: Epinephrine
Drug: Vasopressin
  Arms: Vasopressin

SUMMARY:
Uterine myomas (fibroids or leiomyomas) are the most common benign tumor of the female genital tract and the leading indication for hysterectomy. Although hysterectomy is the definitive treatment of myomas, myomectomy remains the gold standard treatment for women desiring future fertility and uterine conservation3. However, bleeding is often a problem in myomectomy and can results in intraoperative hypovolemic shock, postoperative anemia, pelvic infection, and adhesions with infertility.

A number of interventions have been introduced to reduce hemorrhage during myomectomy. Two categories of interventions can be identified: (a) Vascular interventions on uterine and/or ovarian arteries such as artery clamping, tying, or embolization; (b) pharmacologic interventions such as vasopressin, epinephrine, oxytocin, ergometrine, misoprostol, sulprostone, and gonadotropin-releasing hormone (GnRH) agonist4-11. Of these, intraoperative local injection of vasopressin causing vasospasm is most commonly used. However, there is not a wide consensus on the use of this agent because of serious side effects reported in literature. In addition, in several countries, including France and Italy, vasopressin has not been commercialized because of its potential adverse effects on cardiovascular system.

Epinephrine also induces a vasoconstrictive effect on tissue that lasts longer than that of vasopressin (5-6 hours versus 7-35 minutes) and is used during various gynecological surgeries, endoscopic resection, and dermatologic procedures to reduce blood loss. However, there are a few studies for the use of epinephrine to reduce hemorrhage during myomectomy. Furthermore, a randomized comparison of epinephrine and vasopressin as hemostatic agents during myomectomy has never been conducted. To test the hypothesis that the injections of epinephrine and vasopressin during myomectomy are equivalent in reducing blood loss, the investigators performed this randomized controlled study.

ELIGIBILITY:
Inclusion Criteria:

* women who had myoma-related symptoms such as menorrhagia, pelvic pressure/pain, or infertility
* women who were not pregnant at the time of presentation (i.e., negative for urine pregnancy test or last menstrual period within the last 4 weeks)
* women who were appropriated medical status for laparoscopic surgery (American Society of Anesthesiologists Physical Status classification 1 or 2).

Exclusion Criteria:

* any pelvic abnormalities requiring concomitant surgery
* the presence of pedunculated subserosal or submucosal myoma as a dominant myoma
* the presence of myoma of maximum diameter 10 cm based on the preoperative ultrasound
* more than 4 myomas
* treatment of GnRH agonist or unipristal acetate within 3 months before surgery
* an inability to understand and provide written informed consent.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-05; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Operative blood loss | Surgery date
  The operative blood loss was calculated by the anesthesiology unit as the difference between the total amount of suction and irrigation plus the difference between the total gauze weight before and after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- CHA Gangnam Medical Center, Seoul, South Korea